CLINICAL TRIAL: NCT05348941
Title: Evaluation o Efficacy and Safety of D-chiro-inositol in Insulin Resistant, Obese Patients
Brief Title: Efficacy and Safety of D-chiro-inositol in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DCI_DIET22
Record Dates: First submitted 2022-04-22; First posted 2022-04-27 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Hypocaloric balanced diet
- TECADRIOL (Experimental): Hypocaloric balanced diet plus a food supplement with D-chiro-inositol and alpha-lactalbumin
  Interventions: Dietary Supplement: TECADRIOL

INTERVENTIONS:
Dietary Supplement: TECADRIOL — Food supplement containing an association of D-chiro-inositol and alpha-lactalbumin
  Arms: TECADRIOL

SUMMARY:
The study aims to evaluate the efficacy and tolerability of a food supplement based on D-chiro-inositol in overweight or obese women with insulin resistance, who are approaching a hypocaloric diet

DETAILED DESCRIPTION:
Scientific studies on overweight/obese non-diabetic subjects have shown that weight loss improves insulin sensitivity. In fact, in these subjects weight loss reduces the insulin response to the oral glucose load and lowers plasma concentration of triglycerides.

However, although the insulin value is reduced with diet, it does not reach the levels found in overweight/obese non-insulin resistant subjects.

It has been shown that the supplementation of D-chiro-inositol (DCI), a polyol with an insulin-sensitizing action, can positively affect insulin resistance, avoiding the typical side effects of classic insulin sensitizers. In fact, DCI improves glucose tolerance and increases insulin sensitivity, as demonstrated in hyperinsulinemic women with polycystic ovary syndrome.

Therefore, considering the role of DCI, we want to investigate the efficacy and tolerability of a DCI-based product in overweight / obese women with insulin resistance who are approaching a low-calorie diet.

ELIGIBILITY:
Inclusion Criteria:

* Women between 25 and 40 years old
* Diagnosis of insulin resistance (HOMA ≥2.5)
* 26≤ BMI ≤32

Exclusion Criteria:

* Subjects with no indication for treatment
* Pregnancy and breastfeeding
* Treatment with drugs or supplements that interfere with the mechanism of action of insulin

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
HOMA index | Three time points: change in HOMA index from the baseline to 2 and 4 months
  Reduction of HOMA index

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No